CLINICAL TRIAL: NCT06785441
Title: Older Men's Decision Making About Active Surveillance for Prostate Cancer - Aim 3: Decision Aid Efficacy Testing
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0128
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol describes pilot testing of an educational shared decision-making intervention to help men with localized prostate cancer make decisions with their health care providers about if and when to de-escalate surveillance testing. The project is important because for many patients their cancer does not progress to the point of needed curative treatment or their health status changes such that they are no longer good candidates for treatment. For these men, de-escalating ongoing surveillance (e.g., fewer biopsies or imaging studies) is a reasonable option.

DETAILED DESCRIPTION:
Primary Objective:

The overall goal of this protocol is to test initial efficacy of three versions of an educational tool for use by patients and health-care providers to help men with localized prostate cancer make informed decisions about discontinuation of active surveillance. A pre-post design was selected to provide initial efficacy data of the different versions of the shared decision-making intervention. Thereby, providing preliminary data in preparation for a follow-up comparative study.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Males aged 65 or older
2. Diagnosis of localized prostate cancer
3. Have not received curative intent treatment for their prostate cancer
4. Fluent in English

Care partners/caregivers:

1. Aged 18 or older
2. Fluent in English
3. Involved with the care of an eligible patient (i.e. partner, close friend, family member, companion)

Exclusion Criteria:

Patients

1. Currently receiving treatment for another cancer (primary or recurrence)

Care partners/caregivers

1. None

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Male
Study Population: Male
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2030-02-02 (Estimated)

PRIMARY OUTCOMES:
Preparation for Decision Making Scale | Through study completion and average of 1 year
  The Preparation for Decision Making Scale (PrepDM)19 is a validated scale that assesses whether the decision aid helped prepare a patient to talk with their clinician in making a treatment decision. The scale has 10 items with a 5-point Likert response format,
  Score Scale 1 (not at all) and 5 (a great deal).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lowenstein, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org